CLINICAL TRIAL: NCT05946863
Title: Caudal Anesthesia for Surgical Repair of Fractured Hip or Femoral-neck in Anticoagulated Patients
Brief Title: Caudal Block & Hip Fracture Surgery in Anticoagulated Patient
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Salem2017 Caudal Blk NOF Surg
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hip Fractures; Anticoagulants and Bleeding Disorders
Keywords: Caudal anesthesia
MeSH Terms: conditions — Hip Fractures; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hip fractures are common in elderly patients, and require surgery. Many elderly patients take anticoagulants for vasculopathy treatment. Anticoagulation precludes the use of neuraxial anesthesia because of the risk of epidural bleeding. Caudal anesthesia may be a safe and effective technique in anticoagulated emergency surgical patients.

Quantitative analysis of prospective clinical data. Evaluation of caudal anesthesia efficacy for hip fracture surgery. Analysis of perioperative outcome, and postoperative course.

DETAILED DESCRIPTION:
Hip or femoral neck fractures are common in elderly patients. These fractures require surgical repair. Many elderly patients take regular anticoagulant therapy for vasculopathy. Anticoagulation precludes the use of spinal or epidural anesthesia because of the risk of epidural bleeding. Caudal anesthesia is another form of neuraxial anesthesia that may be safe and effective for hip fracture surgery in anticoagulated elderly patients.

Quantitative analysis of prospective clinical data. It is an evaluation of caudal anesthesia efficacy for hip fracture surgery. This is an analysis of intraoperative analgesia, perioperative outcome, postoperative course, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractured hip or femoral neck who undergo surgical repair

Exclusion Criteria:

* Patients who refuse surgical repair

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult or elderly patients with fractured hip or femoral neck who undergo emergency surgical repair
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 1 month
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandby-Thomas M, Sullivan G, Hall JE. A national survey into the peri-operative anaesthetic management of patients presenting for surgical correction of a fractured neck of femur. Anaesthesia. 2008 Mar;63(3):250-8. doi: 10.1111/j.1365-2044.2007.05328.x. PMID 18289230